CLINICAL TRIAL: NCT00890331
Title: Family Teamwork and Coping Skills Prevention Program
Brief Title: Prevention of Self-care Deterioration in Early Adolescents With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK70917; R01DK070917 (NIH)
Record Dates: First submitted 2009-04-23; First posted 2009-04-29 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes Education (Active Comparator)
  Interventions: Behavioral: Diabetes Education
- TeamWork CS Sessions (Experimental)
  Interventions: Behavioral: TeamWork CS Sessions

INTERVENTIONS:
Behavioral: TeamWork CS Sessions — The intervention focuses on an authoritative parenting approach that emphasizes continued parental involvement in daily disease care. Dyadic coping skills of communication, problem solving, conflict resolution, along with attitude and behavior change are highlighted. Families meet with a study interventionist in conjunction with four consecutive medical appointments.
  Arms: TeamWork CS Sessions
Behavioral: Diabetes Education — Diabetes Education The education comparison group meets with an educational interventionist in conjunction with four consecutive medical appointments. This group focuses on diabetes educational and resource support for parents and their youth with type 1 diabetes.
  Arms: Diabetes Education

SUMMARY:
Establish the efficacy of a brief, clinic-based prevention program of teamwork coping skills for youth and their parents during in a high risk period of early adolescence (11-14 yrs) when parental involvement and self-care deterioration occurs.

DETAILED DESCRIPTION:
Promotion of optimal disease care and metabolic control in youth with Type 1 diabetes is an important goal of disease management during early adolescence. Typically youth assume increasing responsibility for these goals along with parental involvement and guidance. However, as youth progress through adolescence, parents often become less involved in diabetes management and poorer self-care and metabolic control often results.

The goal of the prevention program is to encourage parents to remain involved in their child's diabetes care throughout adolescence and to provide tools to help make that involvement a positive experience. To minimize parent/child conflict that may accompany sustained parental involvement, sessions of the active treatment review the following coping skills: communication, problem solving, conflict resolution, attitude and behavior change. Meetings occur in-clinic in conjunction with four consecutive medical appointments.

The educational comparison group also meets with study researchers for in-clinic sessions that occur in conjunction with four consecutive medical appointments. Families discuss a variety of helpful educational diabetes topics and resources.

The overarching project goal is to demonstrate the efficacy of a brief, prevention focused coping skills program for youth with type 1 diabetes and their parents with the ultimate goal of translation into routine pediatric care.

ELIGIBILITY:
Inclusion Criteria:

* Seen for Diabetes care at Virginia Commonwealth University or Children's National Medical Center
* Child ages 11-14
* Type 1 Diabetes
* Fluent in English
* Ability to comprehend and complete questionnaires independently

Exclusion Criteria:

* The presence of any other major disease
* The presence of any severe diabetic complications which could impair test performance
* Use of any medication that affects the CNS other than insulin
* Inability to speak/comprehend and read English
* Placement in special classes for the mentally disabled

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 2007-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Parental involvement and Disease care behaviors | Baseline, (optional 3, 6, and 9 months) 12, 15, 18 and 24 months

SECONDARY OUTCOMES:
Glycohemoglobin levels, Adverse effects and Blood glucose variability | Baseline, 3, 6, 9, 12, 15, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa S Holmes, Ph.D., Principal Investigator — Virginia Commonwealth University; Randi Streisand, Ph.D., Principal Investigator — Children's National Research Institute; Rusan Chen, Ph.D., Study Director — Georgetown University
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Virginia Commonwealth University, Richmond, Virginia